CLINICAL TRIAL: NCT06356987
Title: Comparison of Laparoscopic Extraperitoneal Closure and Open Herniotomy in Children
Brief Title: Comparison of Laparoscopic Herniotomy and Open Herniotomy in Children
Acronym: Herniotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Muhammad Sharif, PROFESSOR, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0002
Record Dates: First submitted 2024-03-30; First posted 2024-04-10 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Inguinal Hernia
Keywords: Laparoscopic herniotomy; Open herniotomy,; Inguinal Hernia; Children
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: 66 patients with inguinal hernia were randomly divided into two groups (A and B)
Masking Description: 66 patients (33 patients in each group) of laparoscopic extraperitoneal closure and open herniotomy each
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group-A: Laparoscopic hernia repair (Experimental): In group A (33 patients) laparoscopic assisted needle herniotomy was done
  Interventions: Procedure: Herniotomy
- Group B open herniotomy (Active Comparator): In group B(33 patients) open herniotomy was done
  Interventions: Procedure: Herniotomy

INTERVENTIONS:
Procedure: Herniotomy — In Group A Laparoscopic assisted needle herniotomy was done
  Other Names: Laparoscopic herniotomy

SUMMARY:
All patients of age 6 month to 12 years with inguinal hernia were included in study.

Data was collected on detailed proforma regarding age, sex, side ,operative time, cosmesis , and postoperative complications

DETAILED DESCRIPTION:
BACKGROUND: The best method of inguinal hernia repair in children continues to be a topic of debate. Although recent data shows that LPEC is superior and safe but no such data exists in our country. Operative time and recurrence are main concerns. Hence, present study is carried out to compare outcome of LPEC versus OHR in children.

OBJECTIVE: To compare the outcome of laparoscopic percutaneous extra-peritoneal closure and open repair for inguinal hernia in children METHODOLOGY: It was a randomized control trial conducted on 66 patients (33 in each group) presented to our hospital with features of Inguinal Hernia. Patients were admitted after confirmation of diagnosis by ultrasound and complete blood count (CBC) was sent. Pre operatively patients were divided in two groups randomly (Open Hernia Repair group, LPEC group) by closed envelope method. Consent was taken from parents regarding inclusion in the study. All demographic data and results were noted down in a proforma. The collected data was entered and analyzed in computer software SPSS (Statistical Package for Social Sciences) version 26.0.

ELIGIBILITY:
Inclusion Criteria:

All patients of age 6 months to 12 years of either gender having unilateral or bilateral inguinal hernia diagnosed on history, clinical examination and investigations.

Exclusion Criteria:

1. Patients with recurrent inguinal hernia, hydrocele, hernia with undescended testes and Sliding hernia diagnosed on history, clinical examination and investigations.
2. Patients with complicated hernia (e.g. incarcerated ovary), irreducible or obstructed inguinal hernia diagnosed on history, clinical examination and investigations.
3. Patients who cannot tolerate pneumoperitoneum or general anaesthesia.
4. Patients with congenital heart disease, other co-morbid conditions.

   -

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Operative time | 3 months
  Operative time was noted in both groups.
Recurrence | 3 Month
  recurrence was also noted in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sharif, Study Chair — King edward Medical University/Mayo Hospital Lahore
Locations (1):
- Muhammad Sharif, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
plan to share on demand